CLINICAL TRIAL: NCT02204254
Title: Prospective, Open Label, Randomized Study Comparing Bipolar Radiofrequency Potentiated by Infrared Light to Doxycycline in Patient With Papulopustular Rosacea
Brief Title: RosaC-RF : Bipolar Radiofrequency vs Doxycycline in Rosacea
Acronym: Rosac-RF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-AOI-13
Record Dates: First submitted 2014-03-07; First posted 2014-07-30 (Estimated); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea | interventions — Doxycycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radiofrequence (Experimental): 3 sessions of radiofrequency at 3 weeks intervals V1, V2 (W3 or W4) and V3 (between W6 and W8), with clinical examination, evaluation of tolerance, adverse events report, photos, surface biopsy (SSSB), and confocal microscopy (V1 and V3). Follow up visit V4 (M6) with clinical evaluation, photos, SSSB, confocal microscopy, adverse events report and treatment satisfaction.
  Interventions: Device: Radiofrequence
- Doxycycline (Placebo Comparator): doxycycline 100 mg / day for 3 months with clinical evaluation, photos, and confocal SSSB V1 and V4 (M6). Tour V2 M1 for clinical evaluation of safety review, collection of adverse events and issuing end of treatment. Visit V3 M3 on adverse effects.
  Interventions: Drug: Doxycycline

INTERVENTIONS:
Device: Radiofrequence — Associated to arm radiofrequence
  Arms: Radiofrequence
Drug: Doxycycline — doxycycline 100 mg / day for 3 months with clinical evaluation, photos, and confocal SSSB V1 and V4 (M6). Tour V2 M1 for clinical evaluation of safety review, collection of adverse events and issuing end of treatment. Visit V3 M3 on adverse effects.
  Arms: Doxycycline

SUMMARY:
Rosacea is a chronic facial disfiguring dermatosis characterized by different stages like flushing, erythema, telangiectasia and papulo-pustular lesions. Recommended treatments include topical (metronidazole) and systemic (doxycycline) antibiotics with only a suspensive effect. The bipolar radiofrequency (RF) with Elos system (infrared light) is a device emitting an electromagnetic current inducing an increase in temperature when applied on the skin, potentiated by infrared light. The monopolar RF has already been used in rosacea on a small number of cases with positive and prolonged results. RF with Elos system has been evaluated on erythemato-telangiectasic rosacea with encouraging results. Demodex folliculorum (DF) is a long transparent mite which asymptomatically parasitizes pilosebaceous follicle of normal human skin sometimes responsible of inflammatory facial dermatoses. The prevalence and density of DF are increased in rosacea, and DF is suspected to play a role in the pathogenesis of rosacea. DF is sensitive to heat, and the investigators hypothesize that radiofrequency treatment may affect the survival of the mite and should be effective to treat papulopustular rosacea.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be between 18-70 years old
* Subjects with papulopustular rosacea graded moderate to severe (2 or 3) according to the physician global Assessment, and with lesions on the cheeks.
* Prior stop of any topical treatment antibiotic, retinoid, corticoid or other topical treatment for rosacea at least 1 month before the start of the study
* Prior stop of any systemic treatment (antibiotic) two month before the start of the study and for isotretinoin at least 6 months
* Last laser treatment, by lamp, laser or LED, at least 3 months before the start of the study
* Subjects must be abble to lie for more than 30 minutes
* Patient able to understand and sign the informed consent form
* Affiliation to a social security scheme

Exclusion Criteria:

* Women of child bearing/reproductive potential
* Other skin disease or abnormality of the face which could interfere with the evaluation of the different criteria evaluated or with the realization of the RF
* Contraindications to radiofrequency: presence of a defibrillator or pacemaker, dental on the cheeks, dental equipment or metallic orthopedic next to the treated area, skin cancer on the face, progressive systemic disease, uncontrolled hypertension
* Immunosuppression by HIV (determined by examination) or treatment with immunosuppressive
* Tattoos or permanent makeup on the face
* Excessively tanned skin to sunlight, ultraviolet or with tanning creams during the last 2 weeks
* Subject carrying cochlear implants or open wound or in the process of healing
* Minor patient or under tutorship
* Cyanoacrylate or doxycycline allergy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2021-06-07 (Actual)

PRIMARY OUTCOMES:
percent of patients with a score of 0 or 1 severity of rosacea (absent or mild) on a scale of 0-3 (Physician Global Assessment) | at 6 months
  The primary endpoint is the percent of patients with a score of 0 or 1 severity of rosacea (absent or mild) on a scale of 0-3 (Physician Global Assessment) evaluated on photographs by an independent investigator.
  Inflammatory lesions are considered for the evaluation of PGA because it is not expected that the compared treatments improve erythema and telangectasia.

SECONDARY OUTCOMES:
scorecard score | at 6 months
  a) inflammatory lesions count will be assessed on the cheeks. The rate of lesions reduced is the ratio: b ) other symptoms will be achieved by the assessment of erythema (0-3 ) and telangiectasia (score 0-3 ) in the scorecard score.
  c ) The patient satisfaction will be assessed by a Visual Analogue Scale (VAS) .
  d) The evaluation of the density of demodex will be assessed on the skin surface biopsy ( SSSB ) and by confocal microscopy ( MCIV ) e ) The skin temperature during radiofrequency sessions will be reported by infrared thermometer skin temperature during the treatment session RF

CONTACTS AND LOCATIONS:
Overall Officials: Le Duff Florence, Ph, Principal Investigator — CRC, Hôpital Archet, 151 route de saint-antoine de ginestière 06200 Nice
Locations (1):
- CRC, Hôpital de l'Archet, 151 route de saint-ginestière, Nice, Alpes-maritimes, France